CLINICAL TRIAL: NCT05576064
Title: Is Gait Analysis for Proposed Rotational Deformities an Appropriate Use of Resources
Brief Title: Is Gait Analysis for Proposed Rotational Deformities a Useful Resource
Status: Completed | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1 860
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Lower Limb Deformity; Anterior Knee Pain Syndrome; Patellofemoral Pain; Rotation; Deformity
Keywords: Rotational Deformity; Gait Analysis; CT; Patellofemoral Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Congenital Abnormalities | interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Gait analysis — Analysis of gait profile and measures by gait laboratory on patients with suspected lower limb rotational deformities and anterior knee pain
  Other Names: CT

SUMMARY:
Rotational deformities, such as femoral (thigh bone) and tibial (leg bone) torsion, are established causes of patellofemoral (kneecap joint) pain and instability. Currently, computerized tomography (CT) remains the gold standard assessment tool for measuring the degree of rotational deformity. However, there is disagreement as to the thresholds for surgical correction as it is suggested that some individuals compensate for the deformity better than others. Gait (walking) analysis provides important information of the biomechanical parameters undertaken in the knee joint during dynamic movement. In patients with rotational deformities, several variations from normal gait patterns have previously been described by several authors. Therefore, it is questioned whether these parameters can be correlated with the static features of CT scans, in individuals with rotational deformities. This study aims to determine whether gait analysis is a useful tool in the diagnosis and treatment pathway for rotational abnormalities in patellofemoral pain or instability. A secondary aim of this study will be to assess whether gait analysis can detect a rotational deformity in the lower limb and determine whether the changes seen are proportionate to the level of deformity.

Patients to be included in this retrospective study are, adult patients, with presumed rotational deformity of the lower limb, with anterior knee pain, who have been referred to the gait laboratory for assessment, and for CT rotational profiles. Only patients who have given consent to the gait laboratory for their information to be utilised in research will be included. Two researchers will record measures of rotational deformity from the CT images. The gait laboratory assessment includes measurements of biomechanical parameters based on joint movement through the gait cycle - these parameters will be assessed and compared with CT measures for correlation. All research will be conducted at the hospital where the gait laboratory assessment has been performed.

DETAILED DESCRIPTION:
Patellofemoral pain (PFP) is one of the most common disorders in orthopaedic clinics (Rothermich, 2015). The knee pain is said to responsible for 25-40% of annual incidence, though a true prevalence is unknown (Witvrouw, 2014)(Lankhortst et al, 2012). Patient demographics range from young, active individuals to sedentary, elderly individuals (Witvrouw, 2014).

Primary care consultations to orthopaedic and musculoskeletal clinics, from knee pain alone, are reported to account for over 100,000 appointments annually (Smith et al., 2018). This costs the UK economy around £7.4million a year through employment absenteeism, alongside additional costs for non-operative and operative treatment procedures (Smith et al., 2018)(Swan et al., 2010).

Alongside age and activity, an important variable in understanding the epidemiology of PFP is the difference in the incidence and prevalence between genders. Many epidemiologic studies have shown that females have a two-fold higher incidence rate of the disorder than males (Rothermich, 2015).

The aetiology of PFP is evasive and multifactorial. Therefore, patients presenting with this syndrome pose a challenge for the diagnosis and long-term treatment of the pain. An important part of the diagnosis for the disorder is to rule out any other possible causes such as plica syndrome, neuromas or intra-articular pathology (Rothermich, 2015). Combinations of malalignment of the lower extremities, imbalance in muscles of the hips and knee joints, and over use, are the main factors which present most often and are considered causative to the disorder (Rothermich, 2015). One main contributors to PFP is that of lower limb structural factors, such as femoral ante/retro version and tibial torsion (Snow, 2021). These factors are thought to significantly effect gait and muscular function, which results in overloading of the joint and disturbed patellofemoral mechanics (Snow, 2021).

Currently, computerised tomography (CT) is the gold standard tool used to quantify rotational deformity on the lower limb (Snow, 2021). However, CT is a static imaging modality and does not capture the 'real life' dynamic kinetics that occur through movement (Saevarsson et al., 2013). Gait analysis provides important quantitative information of the biomechanical parameters undertaken in the knee joint during dynamic movement. In patients with rotational deformities, these parameters are either heightened or decreased on activity (Arazpour et al., 2016). Therefore, it is questioned as to whether gait analysis can detect a rotational deformity in the lower limb and determine whether the changes seen are proportionate to the level of deformity. Consequently, questioning as to whether gait analysis is an appropriate tool for diagnostic and treatment pathways for PFP.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have previously undergone gait analysis for assessment of patellofemoral pain and or instability
* Have a rotational CT scan available for assessment of femoral and tibial torsion
* Signed research consent form

Exclusion Criteria:

* No available CT scan available
* No gait analysis data available
* No signed gait research consent form

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population will include patients over 16 years of age who have previously had assessment of their gait and who have been diagnosed with suspected rotational deformity and patellofemoral pain/anterior knee pain. All genders will be accepted.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Is gait analysis a useful tool to determine rotational deformity? | 3 months
  The study aims to determine gait analysis is a useful tool in the diagnosis and treatment pathway for rotational abnormalities in patellofemoral pain or instability.

SECONDARY OUTCOMES:
Can gait analysis predict the same rotational deformity as CT | 3 months
  To assess whether gait analysis can detect a rotational deformity in the lower limb and determine whether the changes seen are proportionate to the level of deformity.

CONTACTS AND LOCATIONS:
Overall Officials: Martyn Snow, Principal Investigator — The Robert Jones and Agnes Hunt Orthopaedic Hospital
Locations (1):
- The Robert Jones and Agnes Hunt Orthopaedic Hospital, Oswestry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arazpour M, Bahramian F, Abutorabi A, Nourbakhsh ST, Alidousti A, Aslani H. The Effect of Patellofemoral Pain Syndrome on Gait Parameters: A Literature Review. Arch Bone Jt Surg. 2016 Oct;4(4):298-306. PMID 27847840
- [Background] Lankhorst NE, Bierma-Zeinstra SM, van Middelkoop M. Factors associated with patellofemoral pain syndrome: a systematic review. Br J Sports Med. 2013 Mar;47(4):193-206. doi: 10.1136/bjsports-2011-090369. Epub 2012 Jul 19. PMID 22815424
- [Background] Rothermich MA, Glaviano NR, Li J, Hart JM. Patellofemoral pain: epidemiology, pathophysiology, and treatment options. Clin Sports Med. 2015 Apr;34(2):313-27. doi: 10.1016/j.csm.2014.12.011. Epub 2015 Jan 27. PMID 25818716
- [Background] Saevarsson SK, Romeo CI, Anglin C. Are static and dynamic kinematics comparable after total knee arthroplasty? J Biomech. 2013 Apr 5;46(6):1169-75. doi: 10.1016/j.jbiomech.2013.01.002. Epub 2013 Feb 8. PMID 23394715
- [Background] Smith BE, Selfe J, Thacker D, Hendrick P, Bateman M, Moffatt F, Rathleff MS, Smith TO, Logan P. Incidence and prevalence of patellofemoral pain: A systematic review and meta-analysis. PLoS One. 2018 Jan 11;13(1):e0190892. doi: 10.1371/journal.pone.0190892. eCollection 2018. PMID 29324820
- [Background] Snow M. Tibial Torsion and Patellofemoral Pain and Instability in the Adult Population: Current Concept Review. Curr Rev Musculoskelet Med. 2021 Feb;14(1):67-75. doi: 10.1007/s12178-020-09688-y. Epub 2021 Jan 8. PMID 33420589
- [Background] Tan SS, van Linschoten RL, van Middelkoop M, Koes BW, Bierma-Zeinstra SM, Koopmanschap MA. Cost-utility of exercise therapy in adolescents and young adults suffering from the patellofemoral pain syndrome. Scand J Med Sci Sports. 2010 Aug;20(4):568-79. doi: 10.1111/j.1600-0838.2009.00980.x. Epub 2009 Aug 23. PMID 19706002
- [Background] Witvrouw E, Callaghan MJ, Stefanik JJ, Noehren B, Bazett-Jones DM, Willson JD, Earl-Boehm JE, Davis IS, Powers CM, McConnell J, Crossley KM. Patellofemoral pain: consensus statement from the 3rd International Patellofemoral Pain Research Retreat held in Vancouver, September 2013. Br J Sports Med. 2014 Mar;48(6):411-4. doi: 10.1136/bjsports-2014-093450. No abstract available. PMID 24569145